CLINICAL TRIAL: NCT00411255
Title: Blepharospasm and the Experimental Modulation of Cortical Excitability in Primary and Secondary Motor Areas. A Pilot Study.
Brief Title: Brain Stimulation to Treat Blepharospasm or Meige Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 060192; 06-N-0192
Record Dates: First submitted 2006-12-12; First posted 2006-12-13 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-02-19

CONDITIONS: Blepharospasm; Focal Dystonia
Keywords: Blink Reflex; Transcranial Magnetic Stimulation (TMS); Dystonia; Blepharospasm; BSP; Focal Dystonia
MeSH Terms: conditions — Blepharospasm; Dystonic Disorders; Dystonia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant

INTERVENTIONS:
Procedure: repetitive transcranial magnetic stimulation (rTMS) — Three arms on three different days 180 stimuli will be delivered to the AC with a sham coil, with the H-coil and with a standard circular coil in separate sessions.

SUMMARY:
This research study will examine whether magnetic or electrical stimulation of the brain can improve the involuntary closure of the eyelids in patients with blepharospasm or Meige syndrome; conditions that belong to a group of neurological disorders called dystonias. Blepharospasm and Meige syndrome cause excessive involuntary closure of the eyelids or blinking. In an earlier study of patients with writer's cramp, which is another form of dystonia, symptoms improved temporarily with brain stimulation.

Interested people 18 years of age or older with blepharospasm or Meige syndrome may be eligible for this study. Candidates are screened with a medical history, physical examination and a blink reflex test.

Participants undergo brain stimulation and evaluations before and after the stimulation to test the response, as follows:

Procedures

* Transcranial magnetic stimulation (TMS): A wire coil is held on the patient's scalp. A brief electrical current is passed through the coil, creating a magnetic pulse that stimulates the brain. The subject hears a click and may feel a pulling sensation on the skin under the coil. There may be a twitch in the muscles of the face, arm or leg. The subject may be asked to tense certain muscles slightly or perform other simple actions. The effect of TMS on the muscles is detected with small metal disk electrodes taped to the skin of the arms or legs. TMS is done on eight of the ten test days.
* Repetitive TMS (rTMS): The same procedure as TMS, except repeated magnetic pulses are delivered in short bursts. RTMS is done on eight of the ten test days.
* Theta burst stimulation (TBS): A form of rTMS that involves short bursts of impulses. TBS is done on four study days.
* Cathodal transcranial DC stimulation (tDCS): Two conductive-rubber electrodes placed in saline-soaked sponges are positioned over two areas of the head. A constant weak electrical current flow is applied for 20 minutes. tDCS is done on two study days.

Evaluations

* Physician observation: The subject's eyes are videotaped for 5 minutes before and after each TMS session. A physician then counts how many times the subject blinked during the 5 minutes.
* Questionnaire: Subjects are asked to rate their symptoms before and after brain stimulation.
* Electrophysiological test of the blink reflex: Wires are taped to the skin on the nose and temple to record the eye movement during blinking. A thin plastic rod is placed on the skin over the right e...

DETAILED DESCRIPTION:
BACKGROUND: Blepharospasm (BSP) is a common form of focal dystonia, but the etiology and underlying pathophysiological mechanisms are still obscure. BSP is characterized by excessive involuntary closure of the eyelids. Pathological changes in excitability in the primary motor cortex (MC) and secondary motor areas, such as the anterior cingulate (AC), pre-and supplementary cortex (PMC, SMA) are suggested from electrophysiological and brain imaging studies. It is conceivable that modulation of excitability in some of these areas may lead to amelioration of the symptoms of BSP. Cortical excitability can be experimentally changed by various well-established electrophysiological techniques non-invasively.

METHODS: In this pilot protocol, studying 30 patients with BSP, we will use repetitive transcranial magnetic stimulation (rTMS) over the AC, PMC, SMA and MC in two different inhibitory modes: low frequency rTMS ((lf) rTMS) and continuous theta burst stimulation cTBS. Furthermore, we will apply transcranial direct stimulation (tDCS) in an inhibitory mode (cathodal tDCS) over the MC and low intensity high frequency supraorbital electrical stimulation; the latter will be performed in patients and in 7 healthy subjects. The effects on blepharospasm will be objectively measured by electrophysiological measures (blink reflex recovery curve (BRR), blink rate observation by an investigator blinded to the intervention, and a subjective rating by the patient.

OBJECTIVES: We hypothesize that we will find variable amounts of clinical improvement in BSP patients with these different methods. With this study, we aim to get more insight to the underlying pathophysiological mechanisms of BSP and identify which method of non-invasive brain stimulation may be clinically most efficacious.

ELIGIBILITY:
* INCLUSION CRITERIA PATIENTS:
* Patients with idiopathic BSP or Meige-Syndrome (=BSP plus oromandibular dystonia).
* Age 18 years or older.
* Normal findings in the medical history, physical and neurological examination, except for dystonia (in cases that patients have not had an H& P at the NIH within the last 12 months; they will undergo all these exams on the first study day).
* Last treatment with botulinum toxin more than three months ago.

INCLUSION CRITERIA CONTROLS:

* Age 18 years or older
* Normal findings in the medical history, physical and neurological examination
* No history of neuroleptic medications/ prior use of neuroleptics (such as Haldol(Registered Trademark))
* Not been treated or taken anti-depressants, anti-seizure medication, anticholinergic drugs (such as Artane(Registered Trademark)) and muscle relaxants within the past 4 weeks

EXCLUSION CRITERIA PATIENTS:

Any of the following will exclude a patient from the study:

* Other disease with involuntary blinking (Hemifacial spasm, Tic disorder, Tardive Dyskinesia, Tardive dystonia, etc).
* BSP and normal recovery of R2 in BRR.
* Participation in a clinical trial in the 2 weeks preceding the study.
* History of seizure disorder.
* Pregnancy- a pregnancy test will be performed for women of childbearing potential.
* Symptoms of a clinically relevant illness in the 4 weeks before the first study day, including history of any other neurological disorders or conditions requiring the use of anti-depressants, neuroleptic medications or anti-seizure meds., anticholinergic drugs and muscle relaxants.
* History of neuroleptic medications/prior use of neuroleptics.

EXCLUSION CRITERIA CONTROLS:

A botulinum toxin injection within 3 months of starting the protocol

Any condition that requires the use of anti-depressants, anti-psychotic or anti-seizure medications

Cannot follow the instruction through the entire recording

Not able to provide consent to participate in the study

Patients will be screened and recruited from the outpatient clinic of the HMCS, NINDS. Age matched volunteers will be recruited from the NIH Patient Recruitment and Public Liaison Office.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2006-06-22; Primary Completion 2009-04-07 (Actual); Study Completion 2009-04-07 (Actual)

SECONDARY OUTCOMES:
Patient report the subject rating of their symptoms before and after intervention. | Before, immediately after, and one hour after the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), 9000 Rockville, Bethesda, Maryland, United States

REFERENCES:
- [Background] Antal A, Kincses TZ, Nitsche MA, Bartfai O, Paulus W. Excitability changes induced in the human primary visual cortex by transcranial direct current stimulation: direct electrophysiological evidence. Invest Ophthalmol Vis Sci. 2004 Feb;45(2):702-7. doi: 10.1167/iovs.03-0688. PMID 14744917
- [Background] Aramideh M, Koelman JH, Speelman JD, Ongerboer de Visser B. Eyelid movement disorders and electromyography. Lancet. 2001 Mar 10;357(9258):805-6. doi: 10.1016/s0140-6736(05)71235-6. No abstract available. PMID 11254003
- [Background] Aramideh M, Eekhof JL, Bour LJ, Koelman JH, Speelman JD, Ongerboer de Visser BW. Electromyography and recovery of the blink reflex in involuntary eyelid closure: a comparative study. J Neurol Neurosurg Psychiatry. 1995 Jun;58(6):692-8. doi: 10.1136/jnnp.58.6.692. PMID 7608667